CLINICAL TRIAL: NCT05468047
Title: Effects of a Personal Ketamine-assisted Therapy Experience on Clinicians' Therapeutic Competencies Within a Psychedelic-assisted Therapy Training Program
Brief Title: Ketamine Therapy Experiential Education Study
Acronym: KTEES1
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Psychiatry Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KTEES1
Record Dates: First submitted 2022-07-15; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Psychedelic Experiences; Therapeutic Alliance; Psychology, Perceptual
Keywords: psychedelic-assisted therapy; therapeutic competency; training program; ketamine; mood disorders
MeSH Terms: conditions — Mood Disorders | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This is an observational study following clinicians enrolled in a psychedelic-assisted therapy training program. It will investigate changes in measures of therapeutic efficacy and competency following those who choose to undergo a personal ketamine-assisted therapy experience and those who do not.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine administration (Experimental): These individuals will be provided a personal ketamine-assisted therapy experience as part of an in-person training weekend within a psychedelic-assisted training program.
  Interventions: Drug: Ketamine hydrochloride injection
- No ketamine administration (No Intervention): These individuals will undergo the same psychedelic-assisted training program as those who receive the ketamine experience and will attend the same in-person training weekend; however, these individuals have opted out of ketamine administration by choice or due to contraindication and will not participate in the personal experience.

INTERVENTIONS:
Drug: Ketamine hydrochloride injection — Individuals will be administered a single dose of sub-anesthetic (0.5-0.75 mg/kg; maximum dose of 60 mg regardless of body weight) ketamine hydrochloride injection intramuscularly as part of a ketamine-assisted therapy experience.
  Arms: Ketamine administration

SUMMARY:
This study investigates the use of low-dose (0.5-0.75 mg/kg; maximum dose of 60 mg regardless of body weight) ketamine hydrochloride injection, USP administered intramuscularly to healthy clinicians as part of an experiential learning practice within a psychedelic-assisted therapy (PAT) training program. The primary objective of this study is to test the hypothesis that competencies required for mental healthcare professionals providing PAT are enhanced by undergoing a single ketamine-assisted therapy experience, as part of a PAT training program.

Primary outcomes of this study are self-reported measures of therapeutic efficacy and competency for providing both general and psychedelic-assisted therapy, measured at baseline and four weeks following an academic in-person retreat with optional ketamine administration. Secondary endpoints include measures of personality and magnitude of perceived mystical experiences. Individual changes in scores across time will be calculated, and differences in therapeutic efficacy and competency between clinician trainees who choose to participate in a personal ketamine-assisted therapy session and those who do not will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old
* Are proficient in reading and speaking English
* Competent in decision making capacity
* Enrolled in the IPI Psychedelic Assisted Therapy Training Program
* For those being administered ketamine, able and willing to commit to medication dose, attending all study sessions during the In-Person Experiential Training Weekend, and evaluation instruments
* For those being administered ketamine, willing to refrain from using stimulants, anxiolytics during the day of the study session
* May continue but not change psychiatric medications during the course of the study
* Agree to refrain from using stimulants, anxiolytics during the day of the study sessions
* Agree to refrain from alcohol and marijuana for 24 hours before and the day of study sessions
* Agree to refrain from the use of any psychoactive drug during the course of the study
* Willing to be recorded by video and audio for safety purposes only
* Agree to not operate a car or any other heavy equipment for the rest of the day after the ketamine administration
* If necessary, are willing to be contacted via telephone on a daily basis by the therapist or team after each experiential session
* Able to identify one or two caregiver support persons who can drive participant home, be reached by the team, and provide collateral information as needed
* Willing to inform the investigator within 48 hours if any medical conditions occur or procedures are planned

Exclusion Criteria:

* Unable to provide informed consent
* Anyone currently taking medications contraindicated for ketamine, such as benzodiazepine or lamotrigine
* Anyone deemed at medical screening medically unfit for ketamine exposure including but not limited to:
* prior history of psychotic disorder
* prior history of unstable bipolar disorder
* prior history of personality disorder
* prior history of ketamine use disorder
* active substance use disorder
* untreated migraine headaches
* uncontrolled hypertension
* cardiovascular disease without approval of physician of record
* active or recent suicidal ideation
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Development of Psychotherapists Common Core Questionnaire | 5 weeks
  Scale measuring perceived determinants of professional development as a therapist; this study uses Subscales 8 (21 questions) and 10-1 (1 question) of the DPCCQ. This multi-dimensional measure of therapist development uses questions based on a Likert scale that range from 0 (worst outcome) to 5 (best outcome), -3 (worst outcome) to 3 (best outcome), and 1 (worst outcome) to 6 (best outcome).
Counseling Self Estimate Inventory | 5 weeks
  Scale measuring self-reported measures of general counseling efficacy; Likert scale ranging from 1 (worst outcome) to 6 (best outcome) for each of 37 items.
Psychedelic-Assisted Therapist Self-Efficacy Scale | 5 weeks
  Scale designed to assess psychedelic-assisted therapy-related competencies as defined in the IPI PAT Training Program; Likert scale ranging from 1 (worst outcome) to 5 (best outcome) for each of 45 items.

SECONDARY OUTCOMES:
Big-Five Inventory-2 | 5 weeks
  Self reported personality questionnaire; Likert scale ranging from 1 (worst outcome) to 5 (best outcome) for each of 60 items.
Mystical Experiences Questionnaire | 3 days
  Self-reported scale that assesses ketamine-associated mystical experience and its impact on personal and professional life; Likert scale ranging from 1 (worst outcome) to 5 (best outcome) for each of 30 items.
Columbia Suicide Severity Rating Scale- "Baseline" and "Since Last Visit" versions | 5 weeks
  Self-reported assessment of suicidal ideation and behavior; Yes or No questions assess suicidal ideation and behavior, while Likert scales ranging from 0 (best outcome) to 5 (worst outcome), 1 (best outcome) to 5 (best outcome), or 0 (best outcome) to 2 (worst outcome) for 7 items assess severity.

OTHER OUTCOMES:
Demographic questionnaire | 1 day
  Self-reported baseline demographic information about participants that may be associated with outcomes